CLINICAL TRIAL: NCT01130038
Title: Characteristic of Play: Comparison Between Children With Development Coordination Disorder ( DCD) and Children With Typical Development
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 032/2010k
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Development Coordination Disorder
Keywords: Characteristic of play; DCD; children; Typical Development; Whether there are any differences in the issue of Characteristic of play between Children with DCD and Children with Typical Development
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children with DCD and Typical Development
- Children with DCD: 2 groups Children with DCD and Typical Development

SUMMARY:
There will be found differences in the issue of characteristic of play between Children with Development Coordination Disorder and Children with Typical Development.

ELIGIBILITY:
Inclusion Criteria:

* Children with proper( age expected) intelligence and IQ level
* Study in regular education system
* The DCD diagnosis must be confirmed by a pediatrician

Exclusion Criteria:

* Score above 9 in the Movement Assessment Battery test for Children
* Score below 3.83 in Children Activity Scale for Parents
* routinely take medication
* any physical limitations
* neurologic and/or muscle disease
* any significant hearing and/ or vision limitations

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 4-6 years with Development Coordination Disorder ( DCD) and Children with Typical Development (controlled group)
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clalit Medical Center, Gush Dan (Dan Area), Israel